CLINICAL TRIAL: NCT06513273
Title: Observational GIMEMA Study on the Outcome of Acute Myeloid Leukemia (AML) Patients Treated With New Drugs in Real-life
Brief Title: Observational Study on the Outcome of AML Patients Treated With New Drugs in Real-life (BoxTrial)
Acronym: Box
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: AML2824
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; AML, Adult; Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter, prospective and retrospective observational study aims to evaluate the use and efficacy of new drugs or their combinations in real-life in a population of adult AML patients.

DETAILED DESCRIPTION:
This multicenter, prospective and retrospective observational study (model: case only) aims to evaluate the use and efficacy of new drugs or their combinations in real-life in a population of adult AML patients treated at Italian GIMEMA centers. No additional procedures or visits other than those required by normal clinical practice will be required. every patient will be followed for a minimum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. AML diagnosis according to the ELN guidelines, excluding M3
3. Signed Informed consent, if applicable
4. Treatment initiation with novel drugs in monotherapy or combination, in accordance with the AIFA authorizations, from the AIFA registration up to 31.12.2027 with particular attention to:

   * patients affected by FLT3-mutated AML treated with gilteritinib.
   * patients affected by IDH-mutated AML treated with IDH inhibitors.
   * patients affected by AML in maintenance therapy with oral azacytidine.
   * patients affected by AML treated with glasdegib.
   * patients affected by AML treated with gemtuzumab ozogamicin.
   * other novel drugs or combination for the treatment of AML approved during the study period.

Exclusion Criteria:

Patients included in interventional clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population of adult AML patients treated at Italian GIMEMA centers
Sampling Method: Non-Probability Sample
Enrollment: 397 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
New therapies efficacy in terms of Overall survival | at 24 months
  evaluation of the efficacy of the new therapies or their combinations in the real-life for AML patients in terms of Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Anna Candoni, Principal Investigator — Haematology, University of Modena and Reggio Emilia
Locations (2):
- Italy (2):
  - Ematologia Ente Ecclesiastico Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - UOC Ematologia AOU di SASSARI, Sassari